CLINICAL TRIAL: NCT02276729
Title: A Pilot Randomized Controlled Trial (RCT) of Mirror Box Therapy in Upper Limb Rehabilitation With Sub-acute Stroke Patients
Brief Title: Mirror Box Therapy for Upper Limb Function With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Alison Porter-Armstrong (Other)
Collaborators: Northern Health and Social Care Trust (Other Government)
Responsible Party: Sponsor-Investigator, Dr Alison Porter-Armstrong, Senior Lecturer in Rehabilitation Sciences, University of Ulster
Organization: University of Ulster (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 165094
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Cerebrovascular Accident (CVA); Stroke
Keywords: Upper limb; Rehabilitation; Occupational Therapy; Mirror Box Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirror Box Treatment Group (Experimental): Participants in the intervention group will be required to perform two 20 minute sessions of Mirror Box Therapy, five days/week for the duration of their in-patient stay carried out under the direction of members of the OT stroke team as well as receiving their standard OT treatment for upper limb rehabilitation for the duration of their in-patient stay, which is 3-5 sessions per week of approximately 45 minutes duration. This classic rehabilitation treatment is based upon neurodevelopmental theory using the Bobath approach of postural control and repetitive task training.
  Interventions: Other: Mirror Box Therapy
- Conventional Therapy Control Group (No Intervention): Participants in the control group shall receive their standard OT treatment for upper limb rehabilitation for the duration of their in-patient stay, which is 3-5 sessions per week of approximately 45 minutes duration. This classic rehabilitation treatment is based upon neurodevelopmental theory using the Bobath approach of postural control and repetitive task training.

INTERVENTIONS:
Other: Mirror Box Therapy — Mirror box therapy (MBT) is a relatively new therapeutic intervention that is gaining recognition within OT for the potential it offers in rehabilitation of upper limb function in stroke patients. It is postulated that mirror visual feedback can stimulate neural recovery in the brain using mirrored movements of the non-affected upper limb. It is thought that visual feedback helps recruit dormant motor pathways that replace the damaged pathways and encourage the return of movement to improve upper limb function.
  Arms: Mirror Box Treatment Group

SUMMARY:
Individuals who have sustained a stroke are often left with residual deficits of the upper limb such as impaired movement and sensation. These deficits restrict functional use of the limb in everyday activities and can result in increased dependency upon others to engage in some tasks. Regaining independence through functional use of the arm and hand is an aim of occupational therapy rehabilitation. Mirror box therapy (MBT) is a relatively new innovation being introduced into occupational therapy interventions. Some studies have reported it to be beneficial in upper limb rehabilitation, however, these studies have not involved a sub-acute stroke population. This pilot study aims to provide robust evidence, using RCT design, as to whether this type of therapy may offer greater potential in functional gains in the sub-acute recovery period of stroke than standard rehabilitation of the upper limb alone.

DETAILED DESCRIPTION:
Introduction. Stroke is a major cause of mortality in the United Kingdom with around 111,000 people per year being newly diagnosed. Of the survivors, 50% will be left with significant, long-term effects including residual deficits of the upper limb. Rehabilitation of upper limb impairment rests with the OT who plays a vital role in enabling stroke patients to self-manage their condition and live optimally independent lives. Mirror box therapy (MBT) is a relatively new therapeutic intervention that is gaining recognition within OT for the potential it offers in rehabilitation of upper limb function in stroke patients. Based upon mirror visual feedback originally used in the treatment of phantom limb pain after amputation, neural recovery in the brain can be stimulated using mirrored movements of the non-affected upper limb. It is thought that visual feedback helps recruit dormant motor pathways that replace the damaged pathways and encourage the return of movement, thus mirror box therapy is thought to improve upper limb function through both movement and mental stimulation. However, existing studies are limited due to non- consistent participant post-stroke delay (ranging from 3-12 months). Few studies have included patients in the sub- acute period post stroke (0-3 months), a population considered most likely to benefit from this therapy at the early recovery stage.

Aims and Objectives. The aim of this pilot study is therefore to explore the feasibility of conducting a fully powered randomized controlled trial of mirror box therapy for upper limb rehabilitation within a sub-acute stroke population.

The objectives of the study are to:

1. Evaluate the feasibility of patient recruitment within an in-patient sub-acute single setting;
2. Assess the feasibility of delivering MBT as a component of OT treatment in the sub-acute in-patient population;
3. Evaluate the sensitivity of the outcome measures for use in a fully powered trial and conduct a power calculation;
4. Conduct a preliminary analysis of the data to identify potential treatment gains within and between the 2 groups;
5. Pilot the collection of data to enable cost-consequence analysis to be undertaken as an output of the main RCT.

Sample: 50 participants will be recruited and randomized into two groups (treatment n=25; control n=25) over a 2 year period of 1 January 2015 - 31st Dec 2016.

Sample Size Justification: This sample size will allow us to estimate a standard deviation for the primary outcome, and allow us to estimate participation rate with a precision of +/-12.5% if, as we expect, the rate is in the vicinity of 75%.

Randomization: Block randomization will be undertaken using a computer generated randomization list. Each block is estimated to run over a 16 week period. This will allow for recruitment of between 1-2 new subjects per week and assumes an average inpatient stay of 6 weeks. Group allocation will be concealed in consecutively numbered, opaque sealed envelopes.

Intervention: Participants in both groups shall receive their standard OT treatment for upper limb rehabilitation for the duration of their in-patient stay, which is 3-5 sessions per week of approximately 45 minutes duration. This classic rehabilitation treatment is based upon neurodevelopmental theory using the Bobath approach of postural control and repetitive task training. Participants in the treatment group will be additionally required to perform two 20-minute sessions of mirror box therapy, five days/week for the duration of their in-patient stay. Also based upon neurodevelopmental theory, this treatment creates the illusion of perfect bilateral synchronization of repetitive task training by concealing the affected arm in a mirrored box that reflects the repetitive upper arm movements conducted by the unaffected limb.

Control Group Intervention: Participants will receive standard Occupational Therapy intervention for this population in the sub-acute rehabilitation setting, delivered by members of the OT stroke team. This follows the documented protocol used within the Health and Social Care Trust and progresses through 8 phases from assisted to unassisted movements, gross upper limb movements to wrist and fine finger movement, using remedial and functional activities as well as ward-level rehabilitation.

Treatment Group: Participants in the intervention group will be required to perform two 20 minute sessions of MBT, five days/week for the duration of their in-patient stay carried out under the direction of members of the OT stroke team. Sessions will be conducted at the patient's bedside or in the OT Department. Participants will be seated in a comfortable high chair and positioned in front of an adjustable height table. The mirror box will be positioned on the table in front of the participant. The participant will place or be assisted by the therapist to place the affected arm into the open end section of the nylon box; the mirror section will face the patient's non affected side.

Follow-up data period: We will follow up the initial blocks at both 3 and 6 monthly intervals in order to collect longer term data for use on sustained functional gain as well as for use in economic analysis. We will attempt to follow up as many subjects as possible in the latter blocks at the 3 & 6 monthly intervals.

Analysis: Participation rates to both the complete set of assessments, and to the paired baseline and discharge assessments will be estimated and reported. If compliance to the complete set is similar to compliance with baseline and discharge, then assessment every two weeks will be considered for the main trial. However, if compliance with baseline and discharge falls below 60% this will question the value of conducting a larger study. Differences from baseline at discharge will be analysed using ANCOVA, with baseline assessment as the covariate. The upper 90% limit of the estimated sd will be used in future power calculation. The data from multiple assessments will be analysed using repeated measures ANOVA, and the estimated within and between patient sd used in future calculation. Confidence intervals will be presented for treatment effects, and the upper 95% limits used to inform future planning. The qualitative analysis of the patient exit questionnaire will consist of thematic analysis and synthesis.

Economic Analysis: If the subsequent main RCT demonstrates effectiveness of MBT, then analysis of relative costs and outcomes of the intervention will be demonstrable through a cost-consequence analysis using cost and outcome data gathered through the EQ-5D-5L and information relating to discharge destination and discharge care plans.

Ethics and Data Protection: Ethical approval will be obtained from ORECNI and full research governance approvals before commencement of this project.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over;
* newly admitted inpatient of the rehabilitation ward;
* diagnosis of CVA in the last three months resulting in upper limb motor loss;
* able to follow two part spoken or written commands in the English language;
* upper limb therapy designated as a main portion of goal directed treatment programme;
* consent to take part in the study.

Exclusion Criteria:

* patients who have had a previous CVA
* patients who have gross cognitive impairment
* patients who are unable to understand two part spoken/ written commands in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2018-05-31 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Functional Independence Measure v4 at 6 weeks | Baseline and 6 weeks.
  The FIM/FAM (Version 4) is an 18 item measure of 6 areas of function (self-care; sphincter control; mobility; locomotion; communication and social cognition) grouped into two domains of motor items and cognitive items. Each item is scored on a 7-point likert scale and the score indicates the amount of assistance required to perform each item (ranging from 1 representing total assistance in all areas to 7 representing total independence in all areas), and has been widely used post-stroke18.
Change in Functional Independence Measure v4 at 3 months post-discharge | Baseline and 3 months
  The FIM/FAM (Version 4) is an 18 item measure of 6 areas of function (self-care; sphincter control; mobility; locomotion; communication and social cognition) grouped into two domains of motor items and cognitive items. Each item is scored on a 7-point likert scale and the score indicates the amount of assistance required to perform each item (ranging from 1 representing total assistance in all areas to 7 representing total independence in all areas), and has been widely used post-stroke18.
Change in Functional Independence Measure v4 at 6 months post-discharge | Baseline and 6 months
  The FIM/FAM (Version 4) is an 18 item measure of 6 areas of function (self-care; sphincter control; mobility; locomotion; communication and social cognition) grouped into two domains of motor items and cognitive items. Each item is scored on a 7-point likert scale and the score indicates the amount of assistance required to perform each item (ranging from 1 representing total assistance in all areas to 7 representing total independence in all areas), and has been widely used post-stroke18.

SECONDARY OUTCOMES:
Change in Graded Wolf Motor Function Test (gWMFT) at 6 weeks | Baseline and 6 weeks.
  The gWMFT is a 15-item standardised measure which determines the motor ability of participants by recording functional movement time (0- 120 seconds per item, total = mean of 15 items, maximum score= 120 seconds) and quality of movement (0-7 Likert scale per item with 0= no movement, to 7 = normal movement, total = mean of 15 items, maximum score= 7). This graded version has two levels of each task which can be chosen depending on the participants' general functioning level. The graded version was developed from the original WMFT which has shown to have good reliability and validity. Despite being named a motor assessment, this assessment includes assessment of the upper limb using functional activities and, as such, is considered of relevance to OT outcomes. This outcome measure has also been used by other investigators in previous studies with a stroke cohort.
Change in Graded Wolf Motor Function Test (gWMFT) at 3 months post-discharge | Baseline and 3 months.
  The gWMFT is a 15-item standardised measure which determines the motor ability of participants by recording functional movement time (0- 120 seconds per item, total = mean of 15 items, maximum score= 120 seconds) and quality of movement (0-7 Likert scale per item with 0= no movement, to 7 = normal movement, total = mean of 15 items, maximum score= 7). This graded version has two levels of each task which can be chosen depending on the participants' general functioning level. The graded version was developed from the original WMFT which has shown to have good reliability and validity. Despite being named a motor assessment, this assessment includes assessment of the upper limb using functional activities and, as such, is considered of relevance to OT outcomes. This outcome measure has also been used by other investigators in previous studies with a stroke cohort.
Change in Graded Wolf Motor Function Test (gWMFT) at 6 months post-discharge | Baseline and 6 months.
  The gWMFT is a 15-item standardised measure which determines the motor ability of participants by recording functional movement time (0- 120 seconds per item, total = mean of 15 items, maximum score= 120 seconds) and quality of movement (0-7 Likert scale per item with 0= no movement, to 7 = normal movement, total = mean of 15 items, maximum score= 7). This graded version has two levels of each task which can be chosen depending on the participants' general functioning level. The graded version was developed from the original WMFT which has shown to have good reliability and validity. Despite being named a motor assessment, this assessment includes assessment of the upper limb using functional activities and, as such, is considered of relevance to OT outcomes. This outcome measure has also been used by other investigators in previous studies with a stroke cohort.
Change in EQ-5D-5L15 at 6 weeks | Baseline and 6 weeks.
  The EQ-5D-5L is a widely-used standardized 2 page instrument for use as a measure of health outcome. It is applicable to a wide range of health conditions and treatments and provides a simple descriptive profile of 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) across 5 levels ranging from no problems to extreme problems, and a visual analogue scale of the respondent's self- rated health ranging from 'best imaginable health state' to 'worst imaginable health state'.
Change in EQ-5D-5L15 at 3 months post-discharge | Baseline and 3 months.
  The EQ-5D-5L is a widely-used standardized 2 page instrument for use as a measure of health outcome. It is applicable to a wide range of health conditions and treatments and provides a simple descriptive profile of 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) across 5 levels ranging from no problems to extreme problems, and a visual analogue scale of the respondent's self- rated health ranging from 'best imaginable health state' to 'worst imaginable health state'.
Change in EQ-5D-5L15 at 6 months post-discharge | Baseline and 6 months.
  The EQ-5D-5L is a widely-used standardized 2 page instrument for use as a measure of health outcome. It is applicable to a wide range of health conditions and treatments and provides a simple descriptive profile of 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) across 5 levels ranging from no problems to extreme problems, and a visual analogue scale of the respondent's self- rated health ranging from 'best imaginable health state' to 'worst imaginable health state'.
Change in Canadian Occupational Performance Measure (COPM) at 3 months post-discharge | Baseline and 3 months.
  The COPM is a standardized outcome measure to detect change in a client's self-perception of occupational performance over time. It uses a semi-structured interview format and structured scoring method to detect change scores between assessment and reassessment in everyday occupational activities.
Change in Canadian Occupational Performance Measure (COPM) at 6 months post-discharge | Baseline and 6 months.
  The COPM is a standardized outcome measure to detect change in a client's self-perception of occupational performance over time. It uses a semi-structured interview format and structured scoring method to detect change scores between assessment and reassessment in everyday occupational activities.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Porter-Armstrong, DPhil, Principal Investigator — University of Ulster, Northern Ireland
Locations (1):
- Whiteabbey Hospital, Northern Health and Social Care Trust, Belfast, Co Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scarborough P, Peto V, Bhatnagar P, et al (2009) Stroke Statistics. Dept of Public Health, University of Oxford.
- [Background] Higgins J, Mayo NE, Desrosiers J, Salbach NM, Ahmed S. Upper-limb function and recovery in the acute phase poststroke. J Rehabil Res Dev. 2005 Jan-Feb;42(1):65-76. doi: 10.1682/jrrd.2003.10.0156. PMID 15742251
- [Background] Allied Health Professions Federation (2005). The role of allied health professionals in the treatment and management of people with long term conditions. London: Allied Health Professions Federation
- [Background] Intercollegiate Stroke Working Party (ISWP) (2008), National Clinical Guideline for Stroke. 3rd edition. London, UK: Royal College Physicians
- [Background] Intercollegiate Stroke Working Party (ISWP) (2012). National Clinical Guideline for Stroke. 4th edition. London, UK: Royal College Physicians
- [Background] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Background] Yavuzer G, Selles R, Sezer N, Sutbeyaz S, Bussmann JB, Koseoglu F, Atay MB, Stam HJ. Mirror therapy improves hand function in subacute stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2008 Mar;89(3):393-8. doi: 10.1016/j.apmr.2007.08.162. PMID 18295613
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Stevens JA, Stoykov ME. Using motor imagery in the rehabilitation of hemiparesis. Arch Phys Med Rehabil. 2003 Jul;84(7):1090-2. doi: 10.1016/s0003-9993(03)00042-x. PMID 12881842
- [Background] Uswatte G, Taub E, Morris D, Vignolo M, McCulloch K. Reliability and validity of the upper-extremity Motor Activity Log-14 for measuring real-world arm use. Stroke. 2005 Nov;36(11):2493-6. doi: 10.1161/01.STR.0000185928.90848.2e. Epub 2005 Oct 13. PMID 16224078
- [Background] Dohle C, Pullen J, Nakaten A, Kust J, Rietz C, Karbe H. Mirror therapy promotes recovery from severe hemiparesis: a randomized controlled trial. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):209-17. doi: 10.1177/1545968308324786. Epub 2008 Dec 12. PMID 19074686
- [Background] Morris DM, Uswatte G, Crago JE, Cook EW 3rd, Taub E. The reliability of the wolf motor function test for assessing upper extremity function after stroke. Arch Phys Med Rehabil. 2001 Jun;82(6):750-5. doi: 10.1053/apmr.2001.23183. PMID 11387578
- [Background] Oujamaa L, Relave I, Froger J, Mottet D, Pelissier JY. Rehabilitation of arm function after stroke. Literature review. Ann Phys Rehabil Med. 2009 Apr;52(3):269-93. doi: 10.1016/j.rehab.2008.10.003. Epub 2009 Apr 9. English, French. PMID 19398398
- [Background] Granger CV, Cotter AC, Hamilton BB, Fiedler RC. Functional assessment scales: a study of persons after stroke. Arch Phys Med Rehabil. 1993 Feb;74(2):133-8. PMID 8431095
- [Background] Beninato M, Gill-Body KM, Salles S, Stark PC, Black-Schaffer RM, Stein J. Determination of the minimal clinically important difference in the FIM instrument in patients with stroke. Arch Phys Med Rehabil. 2006 Jan;87(1):32-9. doi: 10.1016/j.apmr.2005.08.130. PMID 16401435
- [Background] Law M, Polatajko H, Pollock N, McColl MA, Carswell A, Baptiste S. Pilot testing of the Canadian Occupational Performance Measure: clinical and measurement issues. Can J Occup Ther. 1994 Oct;61(4):191-7. doi: 10.1177/000841749406100403. PMID 10137673